CLINICAL TRIAL: NCT03835182
Title: Efficacy of Ultrasound Versus Short Wave Diathermy in the Treatment of Lumbar Disc Herniation: a Randomised Control Study
Brief Title: Efficacy of Ultrasound Versus Short Wave Diathermy in the Treatment of a Slipped Disc of the Lower Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Selin Ozen, Physical and Rehabilitation Medicine Specialist, Baskent University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KA13/236
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Radiculopathy; Low Back Pain, Mechanical; Herniated Disk Lumbar
Keywords: lumbar vertebrae; herniated disc; radiculopathy; low back pain; short wave therapy; diathermy; ultrasonic waves
MeSH Terms: conditions — Radiculopathy; Low Back Pain; Intervertebral Disc Displacement; Fever | interventions — Transcutaneous Electric Nerve Stimulation; Exercise Therapy; Control Groups; Exercise

STUDY DESIGN:
Intervention Model Description: Three groups of patients, each containing 31 patients, will be included in the study. Patients in each group will receive a total of ten sessions of physical therapy over a two week period. Each week the patients will receive five sessions of physical therapy on consecutive days. The first group will be treated with a hotpack (20minutes) transcutaneous electrical nerve stimulation applied to the lower back (frequency, ultrasound 1MHz frequency (ten minutes), abdominal and lower back muscle strengthening exercises. The second group will be treated with hotpack, TENS and exercises as previously described plus short wave diathermy at 27.12MHz frequency for ten minutes applied to the lower back. The third group will receive hotpack, TENS applied to the lower back and strengthening exercises as previously described.
Who Masked: Investigator
Masking Description: The investigator assessing the patient before and post treatment will be blind to the treatment received by the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ultrasound group (Active Comparator): Thirty one patients receiving a total of ten sessions of physical therapy over a two week period. Each week the patients will receive five session of physical therapy on consecutive days. The ultrasound group will be treated with a hotpack (20minutes) transcutaneous electrical nerve stimulation (TENS) at a frequency of 100Hz intensity adjusted to the patient's tolerability (twenty minutes) and ultrasound 1MHz frequency (ten minutes) applied to the lower back, abdominal and lower back muscle strengthening exercises.
  Interventions: Device: Ultrasound group
- Short wave diathermy group (Active Comparator): The short wave diathermy group will consist of thirty one patients receiving a total of ten sessions of physical therapy over a two week period. Each week the patients will receive five session of physical therapy on consecutive days. The short wave diathermy group will be treated with a hotpack (20minutes), transcutaneous electrical nerve stimulation (TENS) at a frequency of 100Hz intensity adjusted to the patient's tolerability (twenty minutes) and short wave diathermy at a frequency of 27.12MHz (twenty minutes) applied to the lower back , abdominal and lower back muscle strengthening exercises.
  Interventions: Device: Short wave diathermy group
- Control group (Other): The control group will consist of thirty one patients receiving a total of ten sessions of physical therapy over a two week period. Each week the patients will receive five session of physical therapy on consecutive days. The control group will be treated with a hotpack (20minutes) transcutaneous electrical nerve stimulation (TENS) at a frequency of 100Hz intensity adjusted to the patient's tolerability (twenty minutes) applied to the lower back , abdominal and lower back muscle strengthening exercises.
  Interventions: Other: Control group

INTERVENTIONS:
Device: Ultrasound group — Ultrasound 1 MHz, 1.5 W/cm2 for a total of 10 min applied to the lower back
  Other Names: TENS, hotpack, exercise
  Arms: Ultrasound group
Device: Short wave diathermy group — SWD frequency of 27.12MHz applied in continuous mode (thermic) applied to the lower back for twenty minutes
  Other Names: Curapuls 419 SWD (Enraf-Nonius, Delft, The Netherlands); TENS, hotpack, exercise
  Arms: Short wave diathermy group
Other: Control group — superficial heat, analgesic physical modality and exercise only
  Other Names: TENS, hotpack, exercise
  Arms: Control group

SUMMARY:
Chronic low back pain is a common problem which results in reduced functionality, quality of life and general well being. Conservative treatment includes patient education, exercise, maintaining a healthy body mass index and appropriate modifications to activities of daily living. Physical modalities are used to support the mainstay of treatment and include superficial heat, transcutaneous electrical nerve stimulation (TENS), ultrasound, short wave diathermy , traction, and complimentary therapies.

In the clinical practice of the investigators, diathermy, in the form of ultrasound and short wave, is used to heat deeper tissues, increase tissue elasticity and metabolic rate and reduce pain and muscle spasm. The medical literature to date states that further studies are required to compare the efficacy of different diathermy modalities in the treatment of lower back pain.

The aim of this study was to compare the efficacy of ultrasound to that of short wave diathermy and a treatment program which does not include diathermy in the treatment of a slipped disc.

DETAILED DESCRIPTION:
Chronic lumbar pain is a common problem which results in reduced functionality, quality of life and well being. Chronic low back pain also results in many missed days of work and so is an economic burden as well as a social one. Subacute and chronic conservative treatment of low back pain secondary to a herniated disc of the lower back includes education, lifestyle modifications, and maintenance of a normal body mass index. Physical therapy includes range of motion, strengthening and aerobic exercises alongside use of physical therapy modalities such as superficial heating, low frequency analgesic modalities such as TENS and deep heating modalities such as ultrasonic waves and short wave diathermy.

In Physical Medicine and Rehabilitation departments in Turkey, diathermy is commonly used as an adjunct to exercise in the inpatient treatment of disc herniation of the lumbar region. However, systematic reviews of the effects of diathermy in the form of ultrasound and short wave emphasise the necessity for further studies of their efficacy in the treatment of pain and impact on functionality and quality of life.

Therefore, in this study the investigators aim to compare the efficacy of ultrasound and short wave diathermy in treating pain, improving disability and quality of life in patients with chronic low back pain secondary to disc herniation of the lumbar vertebrae.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age 20-60
* 2)Presenting to the Baskent University Faculty of Medicine Physical Medicine and Rehabilitation Department outpatient clinic
* 3) history of low back pain for greater than three months
* 4) Aetiology of back pain lumbar disc herniation based on history, examination and computed tomography/ magnetic resonance imaging (protruded, extruded disc)

Exclusion Criteria:

* 1)lower extremity neurological deficit, 2) infectious, inflammatory, metabolic, neoplastic, abdominal, pelvic aetiology of back pain. 3) a history of vertebral fracture, spinal surgery, spondylolisthesis 4) heat intolerance/medical contraindication to thermal treatment 5) presence of metal prosthesis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in level of pain | Before treatment, 2 weeks after the commencement of treatment, 6 weeks after the commencement of treatment, 14 weeks after the commencement of treatment
  visual analogue scale (VAS) score from 0 to 10cm for current pain. 0= no pain 10= the worst pain imaginable

SECONDARY OUTCOMES:
Change in level of Disability | Before treatment, 2 weeks after the commencement of treatment, 6 weeks after the commencement of treatment, 14 weeks after the commencement of treatment
  Modified Oswestry Low Back Pain Disability Questionnaire. The Revised Oswestry Disability Index is a condition specific outcome measure for low back pain. The index consists of ten questions with six possible responses regarding the patient's back pain, (scored from 0-5), including the severity of pain and impact on activities of daily living. The minimum obtainable score is 0, the maximum obtainable score is 50. This score is then used to calculate the index percentage using the formula: [total score/(no. of questions answered x 5)]100. The higher the percentage, the greater the level of disability due to low back pain. The minimal detectable change (90% confidence interval)is 10%, change of less than 10% maybe attributed to measurement error.
Change in health related quality of life | Before treatment, 6 weeks after the commencement of treatment, 14 weeks after the commencement of treatment
  Short Form 36 (SF-36).The SF 36 is a generic health survey which assesses health concepts that are pertinent to functional status and well-being such as physical function, bodily pain, role limitations due to emotional and physical problems. The sub scale values are reported: physical functioning, bodily pain, vitality, general health, social functioning, emotional role, physical role, mental health. The lowest and highest possible raw score for the subscales are as follows: physical functioning 10-30, physical role 4- 8, bodily pain 2-12, general health 5-25, vitality 4-24, social functioning 2-10, emotional role 3-6, mental health 5-30. Higher values signify better well being in all subgroups. The raw score is then used to calculate the 'transformed scale: Transformed scale= [(actual raw score- lowest possible raw score)/possible raw score range]100

CONTACTS AND LOCATIONS:
Overall Officials: Sacide N Saracgil Cosar, MD, Study Director — Baskent University Faculty of Medicine
Locations (1):
- Baskent University Faculty of Medicine, Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] Oral A, Ketenci A. Physical Medicine and Rehabilitation Approaches in the Management of Radicular Low Back Pain. A review of the Evidence and Current Recommendations. Turkish Journal of Physlcai and Rehabilitation Medicine 59:57-68, 2013
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Jegede KA, Ndu A, Grauer JN. Contemporary management of symptomatic lumbar disc herniations. Orthop Clin North Am. 2010 Apr;41(2):217-24. doi: 10.1016/j.ocl.2010.01.003. PMID 20399360
- [Background] Fiore P, Panza F, Cassatella G, Russo A, Frisardi V, Solfrizzi V, Ranieri M, Di Teo L, Santamato A. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of low back pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2011 Sep;47(3):367-73. Epub 2011 Jun 8. PMID 21654616
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] Ahmed MS, Shakoor MA, Khan AA. Evaluation of the effects of shortwave diathermy in patients with chronic low back pain. Bangladesh Med Res Counc Bull. 2009 Apr;35(1):18-20. doi: 10.3329/bmrcb.v35i1.2320. PMID 19637541
- [Derived] Ozen S, Guzel S, Senlikci HB, Cosar SNS, Selcuk ES. Efficacy of ultrasound versus short wave diathermy in the treatment of chronic low back pain in patients with lumbar disk herniation: a prospective randomized control study. BMC Sports Sci Med Rehabil. 2023 Nov 20;15(1):157. doi: 10.1186/s13102-023-00769-2. PMID 37986090
- [Derived] Ebadi S, Henschke N, Forogh B, Nakhostin Ansari N, van Tulder MW, Babaei-Ghazani A, Fallah E. Therapeutic ultrasound for chronic low back pain. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD009169. doi: 10.1002/14651858.CD009169.pub3. PMID 32623724